CLINICAL TRIAL: NCT05544565
Title: 3-day Intravenous Antibiotic Treatment Versus 3-day Intravenous Followed by 7-day Oral Antibiotic Treatment for Acute Pyelonephritis in Children 1 Month to 3 Years Old: a Non-inferiority Open Randomized Multicentric Clinical Trial
Brief Title: 3-day IV Antibiotic Treatment Versus 3-day IV Followed by 7-day Oral Antibiotic Treatment for AP in Children
Acronym: PYELOCOURT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP211043; 2021-005627-21 (EudraCT Number)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Pyelonephritis Acute
Keywords: Pyelonephritis acute; Antibiotic therapies; Renal scar; Paediatric
MeSH Terms: interventions — Anti-Bacterial Agents; Defecation

STUDY DESIGN:
Intervention Model Description: Open, multicentric, parallel group non-inferiority clinical trial with 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Discontinuation of treatment (Experimental): For patients randomized in the experimental group, the patient receives 3-day IV therapy and the treatment is interrupted.
  Interventions: Drug: IV Antibacterial Agents; Procedure: Fecal/Rectal Swab; Procedure: PCT assay
- Control group: Usual practice (Other): For patients randomized in the control group, the treatment for acute pyelonephritis is based on the attending clinician's practice and according to the usual practice: 3-day IV therapy followed by a 7-day oral antibiotic therapy.
  Interventions: Drug: IV Antibacterial Agents; Drug: Orally antibacterial agents; Procedure: Fecal/Rectal Swab; Procedure: PCT assay

INTERVENTIONS:
Drug: IV Antibacterial Agents — Ceftriaxone (50 mg/kg once a day by intravenous/intramuscular route) AND/OR Amikacin (20 mg/kg once a day by intravenous/intramuscular route) during 3 days. .
Drug: Orally antibacterial agents — Cotrimoxazole (sulfamethoxazole/trimethoprime) 30mg/kg/day (2 divided doses) OR Cefixime 8mg/kg/day (2 divided doses) during 7 days
  Arms: Control group: Usual practice
Procedure: Fecal/Rectal Swab — Collected by the nurse or the physician (D0,D3,D10 or 17 and D31 or D38), either by a rectal swab, either by fecal swab (dip of the swab in fresh stools < 4 hours, which will occur frequently in our population of children aged 1 month to 3 years, and will in particular be possible for hospitalized children) using a FecalSwabTM, that contains a transport medium.
Procedure: PCT assay — Dosage of procalcitonin (if not performed in standard care) at D0

SUMMARY:
Antibiotic therapies currently recommended for the treatment of acute pyelonephritis (AP) in children, whether fully by the oral route or initially intravenous (IV, 3 days) followed by the oral route, have a duration of 7 to 14 days (10 days in France).

In children with no prior urological malformation, the global clinical and microbiological cure rate after antibiotic treatment completion is around 95%. Recurrence occurs in less than 5% of cases in the 3 months following AP. Renal scarring, when documented, concerns 15% of children 6 months after treatment. Renal scarring can be associated with chronic renal disease.

The investigators hypothesize that 3 days of IV treatment is equivalent to extending to 10 days with an oral to treat AP in children.

The investigators also hypothesize that while achieving equivalent clinical and prevention of re-infections in the following 3 months, 3 days of IV treatment reduces the risk of acquisition of resistant strains of Enterobacteriaceae and increases the gut microbotia diversity compared to extending to 10 days with an oral therapy.

DETAILED DESCRIPTION:
1.0 Hypothesis for the study

Antibiotic therapies currently recommended for the treatment of acute pyelonephritis (AP) in children, whether fully by the oral route or initially intravenous (IV, 3 days) followed by the oral route, have a duration of 7 to 14 days (10 days in France).

In children with no prior urological malformation, the global clinical and microbiological cure rate after antibiotic treatment completion is around 95%. Recurrence occurs in less than 5% of cases in the 3 months following AP. Renal scarring, when documented, concerns 15% of children 6 months after treatment. Renal scarring can be associated with chronic renal disease.

The investigators hypothesize that 3 days of IV treatment is equivalent to extending to 10 days with an oral therapy to prevent long-term renal scarring.

The investigators also hypothesize that while achieving equivalent clinical and microbiological success, and prevention of re-infections in the following 3 months, 3 days of IV treatment reduces the risk of acquisition of resistant strains of Enterobacteriaceae and increases the gut microbotia diversity compared to extending to 10 days with an oral therapy.

2.0 Description of knowledge relating to the condition in question

Acute pyelonephritis (AP) is the most common proven bacterial infection in pediatric clinical practice. It can lead to sepsis or renal abscess and induce long-term complications such as renal scarring. Renal scarring during childhood can lead to hypertension or chronic renal disease at adult age, although the link between AP and chronic renal disease has not been firmly established.

AP is most frequently due to Enterobacteriaceae, mainly Escherichia coli. Extended-spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E) now account for 5% of AP in France and represent a serious threat to public health, owing to limited therapeutic options.

The overall clinical success rate in children treated for AP is around 95% and is not significantly different when ESBL-E are implicated. In children with no prior urological malformation, recurrence in the following 3 months occurs in less than 5% of cases. Antibiotic treatment decreases the risk of renal scarring, which remains important, around 15% (95% CI: 11-18) in the largest meta-analysis. Moreover, delay in treatment of AP is associated with permanent renal scarring.

In children without prior urological malformation, acute complications are exceptional, even in the presence of bacteraemia. Short courses of intravenous (IV) antibiotics (2-4 days) followed by oral therapy have proved to be as efficient as longer courses (7-14 days) of IV treatment. For children aged ≥ 1 month, oral treatment alone for 10 to 14 days has proved non inferior to initial IV antibiotics (2-4 days) followed by oral therapy (total 10 to 14 days).

French Paediatric guidelines recommend a short course (up to 4 days) of IV amikacin and/or ceftriaxone followed by oral therapy (total 10 days), with the possibility, for children aged > 3 months of a 10-day course of oral cefixime [12]. In children initially treated IV, the oral relay occurs once the urine culture and antibiogram are available. The American Association of Pediatrics that focused on children aged 2 to 24 months recommends either an oral or a sequential IV/oral treatment for a total of 7 to 14 days, while the British NICE guidelines recommend an exclusively oral route only for children aged ≥ 3 months

In practice, most centers initiate an IV treatment in a large subset of patients (ongoing practice analysis on the management of AP in children in France, personal data, to be published in 2021). An initial IV treatment is particularly used in young children, with an age cut-off varying between 3 months and 3 years according to the center. It is also used to secure the absorption of the treatment if the child vomits, is unable to take oral antibiotics or is severely unwell.

The excellent short-term and the good long-term clinical outcomes in children treated for AP questions the need for a 10-day course of antibiotics.

In adults, shorter treatments, such as amikacin for 5 days, have been validated for the treatment of uncomplicated AP.

Recently published studies (Zaoutis 2023, Montini 2024) have compared a 5-day oral treatment vs 10-day oral treatment for AP in children. However, the first study (Zaoutis 2023) mainly included (63%) children with a non-febrile urinary tract infection (ie not an AP). The second only included children aged > 3 month. A practice survey conducted prior to our protocol had shown that many departments were already reluctant to treat infants under 1 year old, and particularly those under 3 months old, by oral route, warranting clinical trials including children < 3 month old.

Third-generation cephalosporins (3GC), such as ceftriaxone, rapidly reduce the richness and diversity of the gut microbiota and also select subpopulations of resistant bacteria, particularly by acquisition of extended spectrum beta-lactamases, a major public health issue.

There is no data on the impact of antibiotic relays on the gut microbiota. Since each antibiotic has its own anti-bacterial spectrum, a sequence of treatments could have an additive or even synergistic deleterious effect on the gut microbiota. This may in particular be the case in children treated with IV ceftriaxone for 3 days followed by cotrimoxazole for 7 days, as recommended in France in first intention.

3.0 Summary of relevant pre-clinical experiments and clinical trials

1999 Hoberman et al. Oral versus initial intravenous therapy for urinary tract infections in young febrile children This was a non-inferiority study between oral cefixime for 14 days and intravenous ceftriaxone for 3 days followed by oral cefixime for 11 days. One of the outcomes was the occurrence of renal scarring. It included children aged 1 to 24 months. A total of 306 children were included. Renal scarring at 6 months was noted in 9.8% children treated orally versus 7.2% of children treated intravenously. The study conclude that oral treatment was safe.

The main limit of the study was the lower rate of renal scar in both arms compared to other studies, probably linked to a female/male sex ratio of 9:1 (with a median age of 8 months), when the sex ratio is in favour of boys before 1-year-old.

2007, Montini et al. Antibiotic treatment for pyelonephritis in children: multicentre randomised controlled non-inferiority trial This was a multicentre, randomised controlled, open labelled, parallel group, non-inferiority trial comparing oral co-amoxiclav for 10 days to parenteral ceftriaxone for three days, followed by oral co-amoxiclav for 7 days. Primary outcome was the rate of renal scarring after 12 months. A total of 502 children aged 1 month to <7 years with clinical pyelonephritis were included. Intention to treat analysis showed no significant differences between oral (n=244) and parenteral (n=258) treatment, both in the primary outcome (scarring scintigraphy at 12 months 27/197 (13.7%) v 36/203 (17.7%), and secondary outcomes: time to defervescence, white cell count at day 3, and percentage with sterile urine at day 3 (99.5% n both arms). The results were similar in the subgroups of children older and younger than 2 years (data not shown in the paper).

2012, Boquet et al. Randomized trial of oral versus sequential IV/oral antibiotic for acute pyelonephritis in children PHRC AOM 04 105; NCT00136656 This was a non-inferiority study between oral cefixime for 10 days and IV ceftriaxone for 4 days followed by oral cefixime for 6 days on the occurrence of renal scarring. It included children aged 1 to 36 mont with a first proven urinary tract infection and procalcitonin concentration ≥ 0.5 ng/mL s. The primary endpoint was the proportion of renal scar measured by 99mTc-DMSA renal scintigraphy 6 to 8 months after treatment. The study included a total 171 children of the 698 expected. The incidence of renal scarring was 30.8% in the oral treatment group and 27.3% for children who received the sequential treatment. The trial could not demonstrate statistically the non-inferiority due to insufficient enrolment.

2023, Zaoutis et al. Short-Course Therapy for Urinary Tract Infections in Children: The SCOUT Randomized Clinical Trial PMID: 37358858 ; NCT01595529, This was a randomized clinical noninferiority trial at 2 children's hospitals. Participants included children aged 2 months to 10 years with UTI exhibiting clinical improvement after 5 days of antimicrobials. The study compared another 5 days of antimicrobials (standard-course therapy) or 5 days of placebo (short-course therapy).

The primary outcome, treatment failure, was defined as symptomatic UTI at or before the first follow-up visit (day 11 to 14 A total of 664 children were randomized (639 female [96%]; median age, 4 years): 2 of 328 assigned to standard-course (0.6%) and 14 of 336 assigned to short-course (4.2%) had a treatment failure. There were no differences between groups in rates of UTI after the first follow-up visit, incidence of adverse events, or incidence of gastrointestinal colonization with resistant organisms.

2024, Montini et al. Short Oral Antibiotic Therapy for Pediatric febrile Urinary Tract Infections: A Randomized Trial. [25] PMID: 38146260 This was a multicenter, investigator-initiated, parallel-group, randomized, controlled trial. We randomly assigned children aged 3 months to 5 years with a noncomplicated fUTI to receive amoxicillin-clavulanate for 5 or 10 days.

The primary end point was the recurrence of a urinary tract infection within 30 days after the completion of therapy. Secondary end points were the difference in prevalence of clinical recovery, adverse drug-related events, and resistance to amoxicillin-clavulanic acid and/or to other antibiotics when a recurrent infection occurred.

The study included a total of,175 children and 142 underwent randomization. The recurrence rate of UTI within 30 days of the end of therapy was 2.8% (2/72) in the short group and 14.3% (10/70) in the standard group. The recurrence rate of fUTI within 30 days from the end of therapy was 1.4% (1/72) in the short group and 5.7% (4/70) in the standard group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 month and < 3 years
* For children younger than 3 months, gestational age > 34 WA
* First episode of urinary tract infection
* AP defined by temperature ≥ 38°C on day of diagnosis AND positive urinalysis (white cell counts ≥ 10^4/mL) with a positive urine culture with one Gram- negative bacillus ≥ 104 UFC/mL. The child temperature will have to be measured with a thermometer according to the French national recommendations [Health Insurance website (AMELI ;see: - https://www.ameli. fr/assure/sante/bons-gestes/soins/prendre-temperature); HAS (see: https://www.has-sante. fr/jcms/c_2674284/fr/prise-en-charge-de-la-fievre-chez-l-enfant)].
* Initial treatment by either ceftriaxone AND/OR amikacin
* Outpatient or hospitalised

Non-inclusion Criteria:

* Urine collected by bag
* Urine culture growing more than one dominant bacterium (cf section 6.2 of the protocol)
* Catheter-associated acute pyelonephritis
* Known congenital anomalies of the kidney and genitourinary tract (other than vesicoureteral reflux and pyelocaliceal dilatation < 10 mm)
* Previous surgery of the genitourinary tract (except circumcision in male children)
* Abnormal renal function for age and weight (defined by a serum creatinine >40µmol/L before 1 year and >75µmol between 1 year et 3 years)
* Known immunocompromising condition (e.g., HIV, primary immunodeficiency, sickle cell disease, use of chronic corticosteroids or other immunosuppressive agents)
* Antibiotic prophylaxis for any reason OR antibiotic treatment in the last 7 days (except treatment administered for the AP)
* Known hypersensitivity to at least one of the active substances /excipients: ceftriaxone (including other cephalosporins and other beta-lactams) and amikacin (including other aminoglycosids).
* Known hypersensitivity to at least one of the active substances /excipients: cotrimoxazole (=sulfamethoxazole/trimethoprim) (including other drugs containing sulfonamides) and cefixime (including other cephalosporins)
* Known blood dyscrasias (megaloblastic haematopoiesis)
* Known severe hepatic insufficiency
* Known G6PD deficiency
* No written consent from holders of parental authority
* Non-affiliation to a social security system (as beneficiary or entitled person)
* Children whose follow-up is not carried out in the centre
* Participation in another interventional or minimal risk trial

Randomization criteria :

* Three days of taking antibiotics (IV or IM) (no interruption or discontinuation)
* Positive urine culture with Gram negative bacillus ≥ 10^4 UFC/mL
* Favorable clinical outcome at day of randomization (D2 or D3) defined by temperature < 38°C at day of randomization and absence of fever measured > 38°C for at least 12 hours AND no abdominal pain AND no feeding problem AND investigator agreement
* No renal abscess AND congenital anomalies of the kidney and genitourinary tract (other than vesicoureteral reflux and pyelocaliceal dilatation < 10 mm) on the renal ultrasound performed between D0 and day of randomization
* No more than 1 type of dominant bacteria on the urine culture
* Sensitivity to the initial antibiotic treatment
* Sensitivity to cefixime OR cotrimoxazole

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of febrile urinary tract infection | 28 days (± 3 days) after the completion of antibiotic treatment.
  Demonstrate the non-inferiority of a 3-day intravenous (IV) antibiotic therapy versus a 3-day IV therapy followed by a 7-day oral antibiotic therapy for the treatment of AP in children in term of the is recurrence of febrile urinary tract infection within a 28 -days period after the completion of antibiotic treatment respectively at D31 (+/- 3 days) for the experimental group and D38 (+/- 3 days) for the control group..
  The recurrence will be defined as:
  fever ≥ 38°C associated with a positive urinalysis (white cell counts ≥ 10^4/mL) with a positive urine culture with one Gram-negative bacillus ≥ 10^4 UFC/mL

SECONDARY OUTCOMES:
Clinical cure | D10 (+/- 3 days) for the experimental group and D17 (+/- 3 days) for the control group.
  Demonstrate the non-inferiority of a 3-day IV antibiotic treatment versus a 3-day IV followed by 7-day oral antibiotic treatment for AP in children 1 month to 3 years old in terms of clinical cure, defined by apyrexia AND absence of signs suggestive or urinary infection (abdominal pain, urinary function signs) AND no feeding problem collecting during a medical visit. .
Recurrence of AP | 90 days after the beginning of therapy
  Demonstrate the non-inferiority of a 3-day IV antibiotic treatment versus a 3-day IV/IM followed by 7-day oral antibiotic treatment for AP in children 1 month to 3 years old in terms of recurrence of AP collecting during a phone call.
Colonization with antimicriobial-resistant Enterobacteriaceae | days of randomization and at D10 (+/- 3 days) for the experimental group and D17 (+/- 3 days) for the control group
  Compare between the two treament arms the rate of colonization with antimicrobial-resistant Enterobacteriaceae in the gastrointestinal tract
Bacterial diversity of the intestinal microbiota | Inclusion, randomization and at D10 (+/- 3 days) and D31 (+/- 3 days) for the experimental group, and D17 (+/- 3 days) and D38 (+/- 3 days) for the control group.
  Compare between the two treament arms the bacterial diversity of the intestinal microbiota : alpha-diversity measured by Shannon's index.

CONTACTS AND LOCATIONS:
Overall Officials: Jean GASCHIGNARD, PhD, Principal Investigator — Hôpital Paris-Saclay
Locations (14):
- France (14):
  - CH Sud Francilien, Corbeil-Essonnes, Essonne
  - Paris-Saclay hospital, Orsay, Essonne
  - Antoine Beclère Hospital, Clamart, Haut de Seine
  - Ambroise Paré hospital, Boulogne, Hauts de Seine
  - Children-Teenager hospital, Nantes, Loire Atlantique
  - Jeanne Flandre Hospital, Lille, Nord
  - Robert Debré Hospital, Paris, Paris
  - Meaux Hospital, Meaux, Seine et Marne
  - Jean Verdier Hospital, Bondy, Seine St Denis
  - Intercomunal Créteil Hospital, Créteil, Val de Marne
  - Kremlin Bicêtre Hospital, Le Kremlin-Bicêtre, Val de Marne
  - Andre mignot hospital, Le Chesnay, Yvelines
  - GHEF Site Marne la vallée, Jossigny
  - CHU Toulouse, Toulouse